CLINICAL TRIAL: NCT00500292
Title: A Phase II, Double-blind, Placebo Controlled, Randomized Study to Assess the Efficacy and Safety of 2 Doses of ZD6474 (Vandetanib) in Combination With FOLFOX vs FOLFOX Alone for the Treatment of Colorectal Cancer in Patients Who Have Failed Therapy With an Irinotecan and Fluoropyrimidine Regimen
Brief Title: A Phase II Study of 2 Doses of ZD6474 (Vandetanib) in Combination With FOLFOX vs FOLFOX Alone for the Treatment of Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00047; 2006-005022-23 (EudraCT Number); LPS15025 (Other: Sanofi)
Record Dates: First submitted 2007-07-03; First posted 2007-07-12 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Colorectal; Cancer
Keywords: colorectal; cancer; zactima
MeSH Terms: conditions — Neoplasms | interventions — vandetanib; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): FOLFOX + Placebo vandetanib
  Interventions: Drug: FOLFOX regimen=oxaliplatin, fluorouracil, & folinic acid
- 2 (Experimental): FOLFOX + low dose vandetanib
  Interventions: Drug: Vandetanib; Drug: FOLFOX regimen=oxaliplatin, fluorouracil, & folinic acid
- 3 (Experimental): FOLFOX + high dose vandetanib
  Interventions: Drug: Vandetanib; Drug: FOLFOX regimen=oxaliplatin, fluorouracil, & folinic acid

INTERVENTIONS:
Drug: Vandetanib — once daily oral tablet two dose strengths
  Other Names: AZ6474; ZACTIMA™; SAR390530
  Arms: 2; 3
Drug: FOLFOX regimen=oxaliplatin, fluorouracil, & folinic acid — intravenous infusion

SUMMARY:
The purpose of this study is to determine whether treatment with ZACTIMA (vandetanib) in combination with FOLFOX is more effective than FOLFOX alone for colorectal cancer in patients who have failed therapy with an irinotecan and fluoropyrimidine containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Progression on or following treatment for metastatic colorectal cancer
* Have failed therapy with an irinotecan and fluoropyrimidine containing regimen
* Have World Health Organisation (WHO) performance status 0-2 and life expectancy >12 weeks

Exclusion Criteria:

* Previous treatment with small molecule tyrosine kinase inhibitors of VEGFR or EGFR Prior monoclonal antibodies are permitted, (eg, cetuximab, bevacizumab)
* Previous adjuvant therapy with irinotecan within 12 months of randomisation
* More than one prior course of chemotherapy for treatment of metastatic colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- France (2):
  - Research Site, Lille
  - Research Site, Toulouse
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Poprad
  - Research Site, Trnava
  - Research Site, Žilina
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Hospitalet deLlobregat
  - Research Site, Oviedo
  - Research Site, Santander
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=344&filename=CSR-D4200C00047.pdf
- See also: CSR-D4200C00047.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=344&filename=CSR-D4200C00047.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomised 19 March 2007, last patient randomised 11 Nov 2007, data cut off date 8 March 2008. 109 patients were enrolled in the study.
Pre-assignment Details: 109 patients were enrolled/screened to the study but only 104 patients were entered treatment/randomized.
Groups:
- Vandetanib 100 mg Plus FOLFOX: vandetanib 100 mg plus FOLFOX
- Vandetanib 300 mg Plus FOLFOX: vandetanib 300 mg plus FOLFOX
- Placebo Plus FOLFOX: placebo plus FOLFOX
Period: Overall Study
Arm/Group | Vandetanib 100 mg Plus FOLFOX | Vandetanib 300 mg Plus FOLFOX | Placebo Plus FOLFOX
Started | 32 (randomised patients) | 35 (randomised patients) | 37 (randomised patients)
Completed | 7 (Ongoing study treatment at data cut-off date 8 March 2008.) | 4 (Ongoing study treatment at data cut-off date 8 March 2008.) | 10 (Ongoing study treatment at data cut-off date 8 March 2008.)
Not Completed | 25 | 31 | 27
Not completed — Adverse Event | 3 | 6 | 4
Not completed — Condition under investigation worsened | 21 | 23 | 19
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib 100 mg Plus FOLFOX | Vandetanib 300 mg Plus FOLFOX | Placebo Plus FOLFOX | Total
Number analyzed (Participants) | 32 | 35 | 37 | 104
Age, Continuous [Mean (Full Range); unit: Years] | 57 [34 to 75] | 58 [37 to 71] | 59 [32 to 81] | 58 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 13 | 40
  Male | 16 | 24 | 24 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Objective Disease Progression Event
Description: Number of patients with objective disease progression or death (by any cause in the absence of objective progression)
Time Frame: RECIST tumour assessments carried out at screening and then as per site clinical practice until objective progression. The only additional mandatory tumour assessment visit is at the point of data cut-off (5 March 2008 +/-3 days)
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg Plus FOLFOX | Vandetanib 300 mg Plus FOLFOX | Placebo Plus FOLFOX
Number analyzed (Participants) | 32 | 35 | 37
Participants | 23 | 27 | 24

ADVERSE EVENTS:
Groups:
- Vandetanib 100 mg: vandetanib 100 mg plus FOLFOX
- Vandetanib 300 mg: vandetanib 300 mg plus FOLFOX
- Placebo: placebo plus FOLFOX
Arm/Group | Vandetanib 100 mg | Vandetanib 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/32 | 10/35 | 4/37
Other Adverse Events (participants affected / at risk) | 31/32 | 32/35 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg (N=32) | Vandetanib 300 mg (N=35) | Placebo (N=37)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Device Related Infection (Infections and infestations) | 2 | 0 | 0
Lung Abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 | 0 | 0
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg (N=32) | Vandetanib 300 mg (N=35) | Placebo (N=37)
Leukopenia (Blood and lymphatic system disorders) | 4 | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 13 | 11 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 18 | 13
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Vision Blurred (Eye disorders) | 0 | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 3 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 6 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 16 | 22 | 16
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Gingival Bleeding (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 15 | 24
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 8 | 11 | 10
Toothache (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 9 | 5 | 14
Asthenia (General disorders) | 4 | 8 | 6
Chills (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 8 | 10 | 15
Oedema Peripheral (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 3 | 5 | 9
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 3 | 4 | 5
Bronchitis (Infections and infestations) | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 1 | 0
Electrocardiogram Qt Prolonged (Investigations) | 1 | 6 | 1
Weight Decreased (Investigations) | 3 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 10 | 11 | 9
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2 | 3
Dysaesthesia (Nervous system disorders) | 1 | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 5 | 2
Lethargy (Nervous system disorders) | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 5 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 16 | 12 | 18
Anxiety (Psychiatric disorders) | 0 | 3 | 0
Confusional State (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 3 | 3
Dysuria (Renal and urinary disorders) | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 3
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 3 | 7 | 1
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 7 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 13 | 13 | 5
Phlebitis (Vascular disorders) | 2 | 1 | 1
Phlebitis Superficial (Vascular disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.